CLINICAL TRIAL: NCT02492672
Title: A Multicenter Registry to Evaluate the Long-term Safety and Tolerability of Maintenance Treatment With Iron Sucrose (Venofer) in Pediatric Patients Ages ≥ 2 to ≤ 17 Years With Chronic Kidney Disease
Brief Title: Registry to Evaluate Maintenance Treatment With Venofer in Pediatric Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Registry Protocol
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The current registry is being undertaken to assess the long-term (12 month) safety and tolerability of Venofer in the pediatric population with chronic kidney disease that requires intravenous iron maintenance therapy.

DETAILED DESCRIPTION:
This will be a multicenter, observational, prospective registry collecting long-term (12-month) safety, tolerability, and laboratory data. Subjects will be screened for inclusion criteria if on hemodialysis (HD), peritoneal dialysis (PD) or have non-dialysis dependent (NDD) chronic kidney disease (CKD).

Treatment-emergent adverse events (adverse events starting from the time of the 1st dose of Venofer administered on study) will be collected via site entry of data into a web-based system. Each research investigator will be responsible for entering adverse event information on the appropriate clinical research form as well as reporting such events to the sponsor.

Number of Subjects: 50 evaluable subjects (i.e., took at lease one dose of Venofer and have safety data recorded at the 12 month time point).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 to less than or equal to 17 years
* Subjects must have a diagnosis of either NDD-CKD, PD-CKD or HD-CKD
* Dialysis patients must be on a stable periotoneal (PD) or hemodialysis (HD) regimen for 1 month
* Patient agrees to participate in the registry (i.e., provide adverse event information) for 12 months

Exclusion Criteria:

-

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The current registry is being undertaken to assess the long-term (12 month) safety and tolerability of Venofer in the pediatric population with chronic kidney disease (CKD) that requries intravenous iron maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Treatment- emergent adverse events (TEAE) | 1st Venofer dose through 12 month observation
  Adverse Events starting from from the 1st dose of Venofer adminstered on study through 12 month observation

CONTACTS AND LOCATIONS:
Overall Officials: Linda M. Mundy, MD, PhD, Study Director — American Regent, Inc.
Locations (9):
- United States (9):
  - Stanford University, Palo Alto, California
  - Nemours Orlando A.I. DuPont Hospital for Children, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Medicine, Baltimore, Maryland
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes